CLINICAL TRIAL: NCT00714935
Title: Effects of a Decision Aid for Patients With Coronary Artery Disease on Cardiac Risk Factor Modification Behavior and Health Outcomes
Brief Title: Shared Decision-making: Effects on Cardiac Risk Factor Modification Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Cornelia Ruland, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S-07207a
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease; Decision Making
Keywords: Risk Factors; Risk Reduction Behavior; Counseling
MeSH Terms: conditions — Coronary Artery Disease; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3 (Experimental): Decision Counseling Program(DCP) combined with Coronary Artery Disease Decision Aid (CAD-DA) described in Arm 2
  Interventions: Behavioral: Decision Counseling Program (DCP); Behavioral: Coronary Artery Disease Decision Aid
- 1 (No Intervention)
- 2 (Experimental): Behavioral: Coronary Artery Disease Decision Aid (CAD-DA) presented as a booklet called: "Making Choices: Life Changes to Lower Your Risk of Heart Disease and Stroke"
  The CAD-DA is developed by the Ottawa Health Research Institute and Division of Clinical Epidemiology at Montreal General Hospital, in CAD patients facing the decision of making lifestyle changes to lower their cardiac risk factors and provides patients with information about what they can you do to prevent the disease from progressing.
  Interventions: Behavioral: Coronary Artery Disease Decision Aid

INTERVENTIONS:
Behavioral: Decision Counseling Program (DCP) — An individual decisional counseling program (DCP) to help them comprehend the information, adjust this information to their personal illness history and elicit their preferences for cardiac risk fctor modification behavior in light of this personalized information
  Arms: 3
Behavioral: Coronary Artery Disease Decision Aid — Coronary Artery Disease Decision Aid (CAD-DA) presented as a booklet called: "Making Choices: Life Changes to Lower Your Risk of Heart Disease and Stroke"
  The CAD-DA is developed by the Ottawa Health Research Institute and Division of Clinical Epidemiology at Montreal General Hospital, in CAD patients facing the decision of making lifestyle changes to lower their cardiac risk factors and provides patients with information about what they can you do to prevent the disease from progressing.
  Arms: 2; 3

SUMMARY:
Decision Aids (DA) to inform patients about health care options and help them to participate in their care choices are widely advocated. The main argument for offering patients a choice is that patients' preferences vary, and health professionals cannot always know what is "best" for an individual, specially when different outcomes have different benefits and risk profiles. The standard modes of treatment for patients with coronary artery disease (CAD) are coronary artery bypass graft (CABG) surgery, medication, and angioplasty. All three treatments for CAD work better when combined with cardiac risk factor modification behavior (CRFMB). CRFMB is important for the general public, but it is even more important for people with CAD because people with CAD have more at stake. In this RCT study we will evaluate the effectiveness of a CAD-DA with and witout an additional decision counseling program (DCP) on health outcomes and quality of life to improve enhancement of adherence to cardiac risk modification behavior. The CAD-DA is developed by the Ottawa Health Research Institute and Division of Clinical Epidemiology at Montreal General Hospital, for CAD patients facing the decision of making lifestyle changes to lower their cardiac risk factors. It provides patients with information about what they can you do to prevent the disease from progressing. The DCP is designed to systematically guide patients through the process of deciding what cardiac risk modification behaviors are important for them to carry out. A RCT where 360 CAD patients > 18 of age scheduled for an angiogram at Rikshospitalet University Hospital in Norway (RH) will be randomly assigned to: (1) CAD-DA group where subjects will receive, for take home, the CAD-DA prior to their scheduled angiogram; (2) DCP group where subjects in addition to the CAD-DA will receive an individual decisional counseling program (DCP) from a trained nurse counselor in their homes prior to their angiogram; and (3) the control group who will receive "usual care". Data will be collected at four points: at the initial visit (T1), 2 months (T2), 4 months (T3) and 6 (T4) months after angiogram

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Scheduled for an angiogram
* Able to read, write, and speak Norwegian
* Live within approximately 100 km of Oslo
* Have a telephone

Exclusion Criteria:

- Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life | Repeated measures prior to patients angiogram and 2, 4, and 6 months after angiogram
Health outcomes (angina symptoms, body weight, cholesterol level, blood pressure, health service use) | Repeated measures prior to patients angiogram and 2, 4, and 6 months after angiogram

SECONDARY OUTCOMES:
Intermediate outcome: adherence to cardiac risk factor modification behavior | Repeated measure 2, 4, and 6 months after angiogram
Mediating variables: knowledge, decisional conflict, intention to adhere to cardiac risk factor modification behavior, perceived susceptibility and severity of CAD progression, and benefits and barriers of cardiac risk factor modification behavior | Prior to patients angiogram, and 2 months following angiogram

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia M Ruland, PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Oslo University Hospital, Rikshospitalet,, Oslo
  - Rikshospitalet HF University Hospital, Cardiac Outpatient Clinic, Oslo

REFERENCES:
- [Result] Wensaas L. Effects of a decision aid with and without additional decisional counseling for patients being examined for coronary artery disease on cardiac risk reduction behavior and health outcomes : A randomized controlled trial. Doctoral thesis. University of Oslo, 2012